CLINICAL TRIAL: NCT02781311
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2A Study of Setipiprant Tablets in Androgenetic Alopecia in Males
Brief Title: A Safety and Efficacy Study of Setipiprant Tablets in Androgenetic Alopecia in Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1922-201-002
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Setipiprant (Experimental): Setipiprant 1000 mg (2 X 500 mg) tablets, orally, BID at 12-hour intervals for 24 weeks.
  Interventions: Drug: Setipiprant
- Placebo (Placebo Comparator): Two placebo tablets BID at 12-hour intervals for 24 weeks.
  Interventions: Drug: Placebo
- Finasteride (Active Comparator): Finasteride 1 mg tablet, orally, once daily for 24 weeks.
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Setipiprant — Setipiprant tablets, orally, BID for 24 weeks.
  Other Names: KYTH-105; AGN-241679
  Arms: Setipiprant
Drug: Placebo — Placebo tablets, orally, BID for 24 weeks.
  Arms: Placebo
Drug: Finasteride — Finasteride tablet, orally, once daily for 24 weeks.
  Arms: Finasteride

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of the oral administration of setipiprant tablets 1000 mg twice daily (BID) relative to placebo in 18 to 49 years old males with androgenetic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria:

* Participant has androgenetic alopecia (AGA)
* Participant agrees to maintain current hair care regimen, refraining from hair weaving, hair colorants or dyes and non-study hair growth products during the study.

Exclusion Criteria:

* History of hair loss for reasons other than AGA
* Scarring of the scalp or any condition or disease of the scalp, hair or hair shaft
* Use of products within 6 months of study start used continuously for at least 1 month that could impact hair growth
* Hair-weaving within 6 months
* Use of hair colorants or dyes within 6 months.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Androgenetic Alopecia in Males
Enrollment: 169 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan-En Lin, Study Director — Allergan
Locations (18):
- United States (18):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Petrus Center for Aesthetic Surgery & Hair Transplantation, Little Rock, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - DeNova Research, Chicago, Illinois
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - University of Minnesota Department of Dermatology Division of Clinical research, Minneapolis, Minnesota
  - Wake Forest University Health Sciences Department of Dermatology Medical Center Boulevard, Winston-Salem, North Carolina
  - Cleveland Clinic, Dept of Dermatology, Cleveland, Ohio
  - NW Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Penn State Hershey Medical Center Dermatology Research Office, Hershey, Pennsylvania
  - Radiant Research, Inc., Greer, South Carolina
  - DermResearch, Inc, Austin, Texas
  - Suzzane Bruce and Associates P.A., The Center for Skin Research, Katy, Texas
  - The Education & Research Foundation, Inc, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two placebo tablets, twice daily (BID) at 12-hour intervals for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Setipiprant | Finasteride
Started | 74 | 83 | 12
Safety Population (Treated) | 73 | 81 | 12
mITT Population | 70 | 78 | 11
Completed | 48 | 57 | 8
Not Completed | 26 | 26 | 4
Not completed — Adverse Event | 2 | 6 | 1
Not completed — Withdrawal of Consent | 11 | 12 | 2
Not completed — Lost to Follow-up | 11 | 8 | 1
Not completed — Non-Compliance with Study Drug | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who received study intervention in the study and had a baseline and at least 1 postbaseline measurement for one of the coprimary efficacy measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Setipiprant | Finasteride | Total
Number analyzed (Participants) | 70 | 78 | 11 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (6.08) | 36.3 (6.69) | 34.1 (3.05) | 36.4 (6.25)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 70 | 78 | 11 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59 | 70 | 9 | 138
  Black or African American | 4 | 3 | 0 | 7
  Asian | 4 | 1 | 1 | 6
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Other | 1 | 2 | 0 | 3
  Missing | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 6 | 8 | 0 | 14
  Non-hispanic | 64 | 70 | 11 | 145
Target Area Hair Count (TAHC) Within Left 1 cm^2 Circular Area [Mean (Standard Deviation); unit: terminal hairs/cm^2] — TAHC was measured using digital imaging analysis (macrophotographs) and was reported in terminal hairs/centimeters squared (cm^2). It is a standardized objective quantification of number of hairs within a prespecified target area of scalp at different timepoints. Target area used to count TAHC was 1 cm^2 circular area of clipped hair located at anterior leading edge of vertex thinning area of scalp and centered with a semi-permanent microdot tattoo to ensure same target area was reproduced at each visit. Population: Participants from mITT with data available for analysis at the given timepoint.
  terminal hairs/cm^2
    number analyzed (Participants) | 61 | 70 | 11 | 142
    (all) | 136.7 (55.81) | 148.6 (64.58) | 139.9 (47.72) | 142.8 (59.67)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Target Area Hair Count (TAHC) at Week 24
Description: TAHC was measured using digital imaging analysis and was reported in terminal hairs/centimeters square (cm^2). TAHC is a standardized objective quantification of the number of hairs within a prespecified target area of the scalp at different timepoints, using macrophotography digital images. The total number of terminal hairs (hair width ≥ 30 μm) was calculated from macrophotographs. The target area used to count TAHC was a 1 cm^2 circular area of clipped hair (length approximately 1 mm) located at the anterior leading edge of the vertex thinning area of the scalp and centered with a semi-permanent microdot tattoo to ensure the same target area was reproduced at each visit. A positive change from Baseline indicated improvement (increase in the number of terminal hairs). Missing data are imputed up to Week 24 using last observation carried forward (LOCF) method.
Time Frame: Baseline (Day 1) to Week 24
Population: mITT population included all randomized participants who received study intervention and had a baseline and at least 1 postbaseline measurement for 1 of the coprimary efficacy measures. As per protocol Amendment 1, Finasteride arm group was not included in the analysis model. Number analyzed is participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: terminal hairs/cm^2
Arm/Group | Placebo | Setipiprant
Number analyzed (Participants) | 61 | 70
terminal hairs/cm^2 | 6.7 (3.25) | 7.1 (3.03)
Statistical Analysis 1: Comparison: Placebo vs Setipiprant; Test type: Superiority; p = 0.9239, ANCOVA — P-values were from analysis of covariance (ANCOVA) model including fixed effects of treatment, and covariates of age and baseline TAHC value, with the Type III sum of squares; Least-squares Mean Difference = 0.4, 95% CI 2-sided [-8.38 to 9.23], Standard Error of Mean 4.45

2. Primary Outcome: Subject Self-Assessment (SSA) Score in Hair Growth at Week 24
Description: The SSA consisted of a single-item measure that assesses each participant's perception of change in scalp hair growth. The participant used a standardized global photograph of his scalp taken at the Screening visit presented side by side with a standardized global photograph taken at the postbaseline visit to give a comparative score. The photographs were presented in a blinded and randomized manner to avoid influencing the participant, and response options were on a 7-point ordinal scale (where, -3=Greatly decreased, -2=Moderately decreased, -1=Slightly decreased, 0=No change, +1=Slightly increased, +2=Moderately increased and +3=Greatly increased). The higher the mean SSA value, the more the perception of hair growth from baseline. Missing data are imputed up to Week 24 using LOCF method.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Setipiprant
Number analyzed (Participants) | 68 | 78
score on a scale | -0.2 (0.15) | -0.3 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Setipiprant; Test type: Superiority; p = 0.9101, ANCOVA — P-values were from analysis of covariance (ANCOVA) model including fixed effects of treatment, and covariates of age, with the Type III sum of squares; Least-squares Mean Difference = 0.0, 95% CI 2-sided [-0.42 to 0.37], Standard Error of Mean 0.20

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 8 weeks post last dose (Up to 32 weeks)
Description: Safety population included all the participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Setipiprant | Finasteride
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/81 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/81 | 0/12
Other Adverse Events (participants affected / at risk) | 26/73 | 28/81 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Setipiprant (N=81) | Finasteride (N=12)
Cellulitis (Infections and infestations) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Setipiprant (N=81) | Finasteride (N=12)
Libido decreased (Psychiatric disorders) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 4 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Headache (Nervous system disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0
Influenza (Infections and infestations) | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 3 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0 | 0
Weight increased (Investigations) | 2 | 4 | 0
White blood cell count increased (Investigations) | 3 | 0 | 0
Blood glucose increased (Investigations) | 3 | 0 | 0
Skin abrasion (Immune system disorders) | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Due to change in planned analysis, data of participants in the finasteride arm group were not included in the efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT02781311/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT02781311/SAP_001.pdf